CLINICAL TRIAL: NCT00738361
Title: A Phase 2 Study Of Weekly Infusion Nab-paclitaxel (Paclitaxel Protein-bound Particles for Injectable Suspension) In Patients With Unresectable And Metastatic Uveal Melanoma
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Metastatic Melanoma of the Eye That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Thomas Olencki, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08076; NCI-2011-03176 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Intraocular Melanoma
Keywords: ciliary body and choroid melanoma, medium/large size; iris melanoma; metastatic intraocular melanoma; recurrent intraocular melanoma; extraocular extension melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel (Experimental): Administered via intravenous bolus at a dose of 150 mg/m2 weekly for 3 of 4 weeks every 28 days.
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — 150 mg/m2 weekly for 3 of 4 weeks every 28 days.
  Other Names: Abraxane; paclitaxel protein-bound particles for injectable suspension

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with metastatic melanoma of the eye that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the overall response rate of patients with unresectable, metastatic uveal melanoma treated with paclitaxel albumin-stabilized nanoparticle formulation.

Secondary

* To determine the median progression-free survival of patients treated with this regimen.
* To determine the overall survival of patients treated with this regimen.

OUTLINE: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 8 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed evidence of metastatic/ unresectable uveal melanoma
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension and is ≥10 mm by spiral CT scan
* 18 years or older
* Eastern Cooperative Oncology Group(ECOG)performance status 0, or 1
* No known HIV or Hepatitis B or C
* Patients with brain metastasis are eligible for entry into the study
* Patients must have normal organ/marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelets ≥ 100,000 x 109/L
  * Hemoglobin ≥ 9.0 gm/100 ml
  * Total bilirubin ≤ 1.5. In patients with Gilbert's disease the indirect bilirubin must be less than or equal to 4.0.
  * AST and ALT ≤ 2.5x upper limit of normal
  * Alkaline phosphatase ≤ 2.5x upper limit of normal, unless bone metastases is present in the absence of liver metastasis
  * Creatinine ≤ 1.8 mg/ml or calculated creatinine clearance > 50 mg ml.
  * Calcium <12 mg/dl when corrected for levels of serum albumen
* Patients my have had up to one prior systemic therapy

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering the study or failure to recover from adverse events due to agents administered more than 4 weeks earlier.
* May not be receiving any other simultaneous investigational agents
* No prior malignancy except for adequately treated basal cell cancer, in situ cervical cancer or other cancer for which the patient has been disease free for 2 years.
* Patients who have serious infections or other major uncontrolled medical illnesses.
* Patients who have significant psychiatric illness who in the opinion of the principal investigator would prevent adequate informed consent or render therapy unsafe.
* Patients who are pregnant. Female patients of child bearing potential must have a negative serum pregnancy test and use adequate contraception protection while on study.
* Peripheral neuropathy of > grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Olencki, DO, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-paclitaxel
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- NAb-paclitaxel: Nab-paclitaxel will be administered via intravenous bolus at a dose of 150 mg/m2 weekly for 3 of 4 weeks every 28 days.
Arm/Group | NAb-paclitaxel
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 1 year following last treatment, for a total of approximately 5 years
Measure: Number; unit: patients
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 4
patients | 0

2. Secondary Outcome: Progression-free Survival
Description: Median progression free survival (PFS) in patients with metastatic uveal melanoma who received nab-paclitaxel
Time Frame: up to 1 year following last treatment, for a total of approximately 5 years
Population: all patients progressed at the time of first scan
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 4
months | 6.2 [1.7 to 13.0]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the start of treatment (study day 1) until death to the date of his or her death. If the subject has not died, survival time will be censored on last date the subject was known to be alive.
Time Frame: up to 1 year following last treatment, for a total of approximately 5 years
Measure: Mean (Standard Error); unit: months
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 4
months | 6.1833 (0.8369)

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0 was utilized for Adverse Event (AE) reporting
Arm/Group | NAb-paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAb-paclitaxel (N=4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Constipation (Gastrointestinal disorders) | 2 (3)
Creatinine (Investigations) | 1 (6)
Dermatology Skin (Skin and subcutaneous tissue disorders) | 3 (7) — chest lesion scalp sore mole changes
Diarrhea (Gastrointestinal disorders) | 3 (8)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Edema: limb (General disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 4 (10)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5)
Hemoglobin (Blood and lymphatic system disorders) | 3 (9)
Hemorrhage (Gastrointestinal disorders) | 1 (1) — GI - Varices (rectal)
Hemorrhage (Reproductive system and breast disorders) | 1 (1) — GU - Urinary NOS
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) — Bladder
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2) — Ungual (nails)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (4) — Upper airway NOS
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (27)
Venous insuffiency (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (13)
Alanine Aminotransferase (ALT) (Metabolism and nutrition disorders) | 3 (9)
Aspartate aminotransferase (AST) (Metabolism and nutrition disorders) | 4 (8)
Infection with Normal ANC or Grade 1 or 2 Neutrophils (Infections and infestations) | 1 (2) — Skin (cellulitis)
Infection with normal ANC or Grade 1 or 2 Neutrophils (Infections and infestations) | 1 (2) — Urinary tract NOS and vagina
Nausea (Gastrointestinal disorders) | 3 (6)
Dizziness (Nervous system disorders) | 1 (2)
Sensory Neuropathy (Nervous system disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes